CLINICAL TRIAL: NCT02598414
Title: The Role of Indocyanine Green (ICG) Fluorescence Imaging on Anastomotic Leak and Short-term Outcomes in Robotic Colorectal Surgery: A Prospective Randomized Trial
Brief Title: The Role of Indocyanine Green (ICG) Fluorescence Imaging on Anastomotic Leak in Robotic Colorectal Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Collaborators: Acibadem Atakent University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICG-COLORECTAL
Record Dates: First submitted 2015-11-02; First posted 2015-11-05 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Colon Neoplasms; Rectal Neoplasms; Inflammatory Bowel Disease; Diverticular Disease
Keywords: Colorectal Disease; Robotic Surgery; Indocyanine Green Fluorescence Imaging; Anastomotic Leak; Short-term Outcomes
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Inflammatory Bowel Diseases; Diverticular Diseases; Anastomotic Leak | interventions — Indocyanine Green

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bowel Anastomosis Under ICG Guidance (Experimental): Patients undergo robotic colon/rectal resection and anastomosis with near-infrared ICG fluorescence imaging.
  Interventions: Procedure: Near-infrared ICG fluorescence imaging; Device: FireFly™
- Standard Bowel Anastomosis (Active Comparator): Patients undergo robotic colon/rectal resection and anastomosis without near-infrared ICG fluorescence imaging.
  Interventions: Procedure: Traditional bowel anastomosis

INTERVENTIONS:
Procedure: Near-infrared ICG fluorescence imaging — Patient will have their bowel anastomosis assessed intraoperatively by near-infrared technology after indocyanine green has been injected intravenously at a concentration of 2.5 mg/ml. This procedure will be repeated twice during surgery, the first time before and the second time after the anastomosis has been done. The microvascularization at the anastomosis site will be assessed using a robotic fluorescence imaging device (FireFly™).
  Other Names: Near-infrared fluorescence imaging; Indocyanine green
  Arms: Bowel Anastomosis Under ICG Guidance
Procedure: Traditional bowel anastomosis — Traditional bowel anastomosis will be performed without ICG fluorescence imaging.
  Arms: Standard Bowel Anastomosis
Device: FireFly™ — The microvascularization at the anastomosis site will be assessed using a robotic fluorescence imaging device (FireFly™).
  Arms: Bowel Anastomosis Under ICG Guidance

SUMMARY:
In colorectal surgery, anastomotic leak and its septic consequences still remain as the most concerning complications resulting in substantial morbidity and mortality. A common determining factor for assessing the viability of a bowel anastomosis is adequate arterial perfusion to ensure sufficient local tissue oxygenation. Intraoperative near-infrared fluorescence (INIF) imaging using indocyanine green (ICG) dye is a novel technique which allows the surgeon to choose the point of transection at an optimally perfused area before creating a bowel anastomosis. Recently, the INIF imaging system has been installed on the robotic systems and this helps identify intravascular NIF signals in real time.

Although reports from several case series and retrospective cohorts have described the feasibility and safety of this imaging system during robotic colorectal surgery, to date, no studies have addressed more systematically the outcomes of this technique in robotic surgery. Considering the limitations of these reports, investigators aim to conduct a prospective randomized trial to compare robotic procedures with or without INIF imaging in patients undergoing colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to give informed consent for participation in the study
* Subject is willing and able to comply with the study procedures
* Subject is diagnosed with colon/rectal neoplasia, inflammatory bowel disease, diverticular disease requiring surgical excision
* Subject is scheduled for robotic colon or rectal resection
* A negative pregnancy test for women of childbearing potential prior to surgery

Exclusion Criteria:

* Subjects present with bowel obstruction or perforation
* Subject undergo emergency surgery
* Subject with ASA IV, V
* History of allergy or hypersensitivity against indocyanine green
* Pregnant or breast-feeding women
* Subject has uremia (serum creatinine >2.5 mg/dl)
* Subject is undergoing palliative surgery or who is terminally ill
* Subject who is unable to discontinue warfarin anticoagulation 5 days before surgery
* Subject taking phenobarbital, phenylbutazone, primidone, phenytoin, haloperidol, nitrofurantoin, probenecid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak rate | Postoperative 30 days
  Anastomotic leak rate within 30 post operative days

SECONDARY OUTCOMES:
Complication rate | Postoperative 30 days
  Complication rate within postoperative 30 days
Mortality | Postoperative 30 days
  Mortality within 30 post operative days

CONTACTS AND LOCATIONS:
Overall Officials: Bilgi Baca, MD,Prof.Dr., Principal Investigator — Department of General Surgery, Acibadem University, Atakent Hospital
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Ris F, Hompes R, Cunningham C, Lindsey I, Guy R, Jones O, George B, Cahill RA, Mortensen NJ. Near-infrared (NIR) perfusion angiography in minimally invasive colorectal surgery. Surg Endosc. 2014 Jul;28(7):2221-6. doi: 10.1007/s00464-014-3432-y. Epub 2014 Feb 25. PMID 24566744
- [Result] Jafari MD, Wexner SD, Martz JE, McLemore EC, Margolin DA, Sherwinter DA, Lee SW, Senagore AJ, Phelan MJ, Stamos MJ. Perfusion assessment in laparoscopic left-sided/anterior resection (PILLAR II): a multi-institutional study. J Am Coll Surg. 2015 Jan;220(1):82-92.e1. doi: 10.1016/j.jamcollsurg.2014.09.015. Epub 2014 Sep 28. PMID 25451666